CLINICAL TRIAL: NCT04492761
Title: Family Impact of Polyhandicap: Mixed Methodological Approach
Brief Title: Family Impact of Polyhandicap: a Mixed Methodological Approach
Acronym: PolyMiMe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-53
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Polyhandicap

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: qualitative study — The qualitative approach will be based on content analysis of - Isemi-structured nterviews of families

SUMMARY:
Polyhandicap (PLH) is a complex disability condition corresponding to a chronic affliction occurring in an immature brain, leading to the combination of profound mental retardation and serious motor deficit, resulting in an extreme restriction of autonomy and communication. In a preliminary work, we demonstrated that French families reporteda deterioration of the quality of life. This first study, based on a cross-sectional study and quantitative methods, did not allow to explore: 1) the dynamic aspect and the evolution over time of this experience, 2) the mechanisms underlying the difficulties encountered, the needs and expectations of families

ELIGIBILITY:
Inclusion Criteria:

* Familial caregivers: member of a family of a polyhandicapped person aged from 8 to 35 years old
* Patients: with severe polyhandicap defined by the combination of motor deficiency and intellectual impairment associated with everyday life dependence, restricted mobility and age at onset of cerebral lesion below 3 years old
* Written consent signed by caregivers for participation

Exclusion Criteria:

* caregivers refusing to participate

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - family member (parent, siblings, uncle / aunt) of a person with a severe multiple disability whose age is between 8 and 35 years old
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Qualite of life | 5 years
  WHOQOL-Bref

SECONDARY OUTCOMES:
interview content | 2 hours
  semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Jean Olivier ARNAUD, Study Director — Assistance Publique Hôpitauix de Marseille
Locations (1):
- Assistance Publique Hôpiatuix de Marseille, Marseille, France